CLINICAL TRIAL: NCT01173068
Title: A Prospective Observational Study of Ertapenem in Outpatient Parenteral Antibiotic Therapy (OPAT) for Complicated Urinary Tract Infections.
Brief Title: An Observational Study of Ertapenem in Outpatient Parenteral Antibiotic Therapy (OPAT) for Complicated Urinary Tract Infections.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Medicine, A/Prof Dale Fisher, National University Hospital, Singapore
Other Study IDs: DSRB Domain E/10/312
Record Dates: First submitted 2010-07-28; First posted 2010-07-30 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Urinary Tract Infections
Keywords: Ertapenem; Clinical outcome; Complicated Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections | interventions — Ertapenem

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Ertapenem — Prescribed IV Ertapenem 1gm (or renally adjusted dose) will be administered every 24 hours. The duration of treatment will be determined by the clinician and this typically is 2 weeks, or as clinically indicated.
  Other Names: Invanz

SUMMARY:
The aim of this study is to determine the outcomes when using ertapenem for complicated urinary tract infections in the OPAt setting.

The study hypothesis: Ertapenem is an efficacious and safe therapeutic option for complicated urinary tract infections in the OPAt setting.

DETAILED DESCRIPTION:
Enterobactericae spp. is a common cause of urinary tract infections. The prevalence of quinolone-resistance in Enterobactericae is rising and often co-exists with expression of extended-spectrum beta-lactamases (ESBL, limiting viable outpatient therapeutics options.

In Singapore, there is an increasing trend of treating patients who respond favourably to initial antimicrobial therapy in the outpatient setting (Fisher, et.al, 2006). Ertapenem is one of several agents with excellent antimicrobial activity against Enterobactericae (including ESBL producers). In view of its safety profile and its viability in elastromeric pump, it has great potential to be used in OPAT patients.

There is no study analyzing outcomes in a large cohort of patients with complicated urinary tract infections treated with ertapenem.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 21 years old to 70 years old.
* Diagnosed with complicated urinary tract infection due to pathogen susceptible to ertapenem based on microbiology report, and the use of ertapenem is deemed clinically appropriate by the Infectious Disease physician in charge.

Exclusion Criteria:

* Hypersensitivity reactions to Ertapenem.
* Participation in another interventional clinical investigation within 30days
* Unable to obtain informed consent.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults OPAT patients diagnosed with complicated urinary tract infections and whom require IV Ertapenem will be enrolled over a period of 1-2 years.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-08; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcome | within 14 days of treatment and within 1 months after the treatment completion.
  Measured by:
  1. Clinical features within 14 days of treatmnet:(improving/resolving/deteriorating) during therapy in OPAT eg dysuria,suprapubic pain, frequency, fever, urinalysis.
  2. Clinical features of recurrences with 1 month after therapy completion
  3. Presence of hospitalization and/or
  4. Mortality

SECONDARY OUTCOMES:
Microbiology outcome | 30 days after completion of treatment
  Measured by:
  urine culture results at the end of treatment and 30 days subsequent

CONTACTS AND LOCATIONS:
Overall Officials: Dale A Fisher, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Brink AJ, Richards GA, Schillack V, Kiem S, Schentag J. Pharmacokinetics of once-daily dosing of ertapenem in critically ill patients with severe sepsis. Int J Antimicrob Agents. 2009 May;33(5):432-6. doi: 10.1016/j.ijantimicag.2008.10.005. Epub 2008 Dec 16. PMID 19091521
- [Background] Fisher DA, Kurup A, Lye D, Tambyah PA, Sulaiman Z, Poon EY, Lee W, Kaur V, Lim PL. Outpatient parenteral antibiotic therapy in Singapore. Int J Antimicrob Agents. 2006 Dec;28(6):545-50. doi: 10.1016/j.ijantimicag.2006.08.018. Epub 2006 Nov 13. PMID 17097856
- [Background] Teng CP, Chen HH, Chan J, Lye DC. Ertapenem for the treatment of extended-spectrum beta-lactamase-producing Gram-negative bacterial infections. Int J Antimicrob Agents. 2007 Oct;30(4):356-9. doi: 10.1016/j.ijantimicag.2007.05.016. Epub 2007 Jul 13. PMID 17631986